CLINICAL TRIAL: NCT00001539
Title: A Comprehensive Clinical, Microbiological and Immunological Assessment of Patients With Suspected Post Treatment Lyme Disease Syndrome and Selected Control Populations
Status: Recruiting | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 960052; 96-I-0052
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2025-11-19 (Actual); Status verified 2025-11-06

CONDITIONS: Lyme Disease
Keywords: Borrelia Burgdorferi; Lyme Borreliosis; Tick-Borne Disease; Natural History; Lyme Disease
MeSH Terms: conditions — Lyme Disease; Tick-Borne Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (8):
- healthy volunteers: healthy individuals who have never had Lyme disease
- Lyme arthritis: patients with suspected Lyme arthritis
- multiple sclerosis controls: patients diagnosed with multiple sclerosis who have never been diagnosed with Lyme disease
- OspA vaccine: patients who received two doses of the OspA vaccine
- PTLDS: presumed PTLDS
- PTLDS for screening: patients suspected of PTLDS for screening
- recovered controls: patients who were diagnosed with Lyme disease, treated, and fully recovered
- seropositive controls: patients who are seropositive for Lyme disease, but have no manifestations/symptoms and have never been treated for Lyme disease

SUMMARY:
This study will determine whether patients who have been infected with the Lyme bacteria, Borrelia burgdorferi, and treated with antibiotics still have the bacteria alive inside them and whether it is causing their symptoms. The information from this study may serve as a basis for developing stringent diagnostic criteria for Lyme disease and the establishment of future treatment trials.

Individuals in the following categories may be eligible for this study: chronic Lyme disease; chronic Lyme arthritis; seropositive control (are infected with the bacteria that causes Lyme disease but do not have disease symptoms); recovered control (have been sick with Lyme disease but were treated successfully and are currently well); control with multiple sclerosis (patients with multiple sclerosis); and healthy volunteers. Patients in the chronic Lyme disease category must be age 13 and above; all others must be age18 and above. Candidates will be screened with blood and urine tests.

Participants will have a physical examination and the following tests:

Blood tests Includes HLA-typing, a genetic test of immune system markers;

Leukapheresis Collection of large numbers of white blood cells Whole blood is collected through a needle in an arm vein. The blood circulates through a machine that separates it into its components. The white cells are removed and the rest of the blood is returned to the body, either through the same needle used to draw the blood or through another needle in the other arm. (Alternatively, patients will 100 cc (about 7 tablespoons) of blood drawn.);

Lumbar puncture (spinal tap) Collection of cerebrospinal fluid (CSF, fluid that bathes the brain and spinal cord). A local anesthetic is administered and a needle is inserted in the space between the bones in the lower back where the cerebrospinal fluid circulates below the spinal cord. A small amount of fluid is collected through the needle;

Magnetic resonance imaging (MRI) of the brain Imaging of the brain using a strong magnetic field and radio waves instead of X-rays. During the scan, the patient lies on a table in a narrow cylinder containing a magnetic field. He or she can speak with a staff member via an intercom at all times during the procedure;

Neuropsychologic testing;

Some participants may also have a hearing test and urine collection.

Participants whose test results are positive for Borrelia burgdorferi will be followed at NIH at intervals of 3 to 6 months until it is determined whether there is infection. Those who are infected will be offered treatment with the antibiotic ceftriaxone. Following treatment, patients will return to the NIH Clinical Center for follow-up visits 1 week after treatment and again at 3, 6 and 12 months. The lumbar puncture, hearing examination, blood and urine tests will be repeated at these visits to evaluate the response to treatment, and the leukapheresis will be repeated for research purposes. Patients whose MRI was abnormal during therapy will have a repeat MRI at the 3-month, 6-month and 1-year visits.

All participants with chronic Lyme disease, chronic Lyme arthritis, seropositive controls and recovered controls may be reevaluated at intervals of 6 to 12 months.

DETAILED DESCRIPTION:
Lyme disease has emerged as the leading vector-borne disease in the United States. Despite how much has been learned about Lyme borreliosis in the past decade, there are still many remaining areas of uncertainty. One fundamental question is whether persistent signs and symptoms of disease, despite the administration of what is currently considered to be adequate antibiotic therapy, are due to ongoing active borrelial infection, to a post-infectious syndrome, to irreversible sequelae of earlier tissue injury or due to a condition unrelated to Lyme disease. Reliable objective markers of infection, of clinical status and of host responses to the organism are required to discern the scope and the implications of persistent borrelial infection, the effectiveness of current treatment options, and the development of new therapeutic approaches. The goal of this study is to assemble and follow a well-characterized cohort of patients with post-treatment Lyme disease syndrome and relevant controls that will yield a prospective database upon which stringent diagnostic criteria can be established and future therapeutic trials can be designed.

ELIGIBILITY:
* INCLUSION CRITERIA:

SCREENING FOR SUSPECTED PTLDS

Age >= 13 years old, suspect of suffering from Lyme disease

POST-TREATMENT LYME DISEASE SYNDROME (PTLDS)

For the purposes of this study, PTLDS is defined as (1) occurring in male or female patients aged 13 and above (2) who have been diagnosed with confirmed or probable Lyme disease per CDC definition (https://wwwn.cdc.gov/nndss/conditions/lyme-disease/case-definition/2017/). Study physician will review history to confirm probable cases. (3) They have received recommended antibiotic therapy (4) and have persistent or relapsing symptoms and/or signs for at least six months after therapy [4, 5]. (5) They also should have no other documented explanation for their signs and symptoms.

LYME ARTHRITIS CONTROLS

For the purposes of this study, Lyme arthritis is defined as occurring in an otherwise healthy male or female aged 18 and above who have intermittent episodes of arthritis involving one or few joints, without any other cause being documented, and have positive serum antibodies to B. burgdorferi confirmed by IgG Western blot according to the CDC criteria.

RECOVERED CONTROLS

For the purposes of this study, a recovered control is defined as an otherwise healthy male or female aged 18 and above who has had confirmed or probable Lyme disease, fulfilling the CDC Lyme Disease National Surveillance Case Definition (appendix 5), and who had received accepted antibiotic treatment for Lyme disease [5] (at least 3 months since the end of antibiotic therapy before protocol evaluation) and who are currently asymptomatic.

SEROPOSITIVE CONTROLS

For the purposes of this study, a seropositive control is defined as an otherwise healthy male or female aged 18 and above who has positive serum IgG antibody response to B. burgdorferi by Western blot according to the CDC criteria and are asymptomatic and who recall no episodes of disease compatible with Lyme infection and have not received antibiotic therapy for Lyme

disease.

OSPA VACCINATED CONTROL

For the purposes of this study, an OspA vaccinated control is defined as an otherwise healthy male or female age 18 and above who has received at least two doses of the OspA vaccine for Lyme disease (Lymerix ). These controls may have a positive ELISA for B. burgdorferi but a negative (or unreadable) IgG western blot.

MULTIPLE SCLEROSIS CONTROLS

For the purposes of this study, a multiple sclerosis control is defined as an otherwise healthy male or female aged 18 and above with relapsing-remitting or progressive multiple sclerosis as defined by the Clinical Trial Committee of the National Multiple Sclerosis Society and no evidence of prior exposure to B. burgdorferi as indicate by negative history for Lyme disease and negative western blot for B. burgdorferi in the serum by the CDC criteria. Patients should have a Kurtzke or Expanded Disability Status Scale (EDSS) between 1 and 5.

HEALTHY VOLUNTEERS

For the purpose of this study, a healthy volunteer is defined as healthy male or female, age 18 and above, with no history compatible with Lyme disease and negative serological testing to B. burgdorferi by the CDC criteria.

GENERAL EXCLUSION CRITERIA

1. Age less than 18 (less than 13 for patients with PTLDS)
2. Weight less than 70 Lb. (35 kg)
3. Pregnancy or lactation
4. Women with childbearing potential who are sexually active with a male partner and unwilling to use effective contraception during the evaluation and treatment phases of the protocol.
5. Clinically significant laboratory abnormalities including positive test for syphilis (RPR), HBsAg, anti-HCV, anti-HIV.
6. Chronic medication use will be evaluated in a case-by-case basis.
7. Not able to understand all of the requirements of the study or unable to give informed consent and/or comply with all aspects of the evaluation.
8. All study participants must agree to allow their samples to be used for future research.

EXCLUSION CRITERIA FOR PTLDS PATIENTS AND LYME ARTHRITIS CONTROLS:

In addition to the general exclusion criteria, these individuals will be excluded for:

1. Use of immunosuppressive drugs such as systemic (but not topical or inhalant) steroids and cytotoxic agents.
2. History of any recognized autoimmune disease such as rheumatoid arthritis, vasculitis, systemic erythematous lupus, etc.
3. Serious pre-existing or concurrent chronic medical or psychiatric illnesses other than Lyme disease.
4. Past history of significant head trauma, alcohol or substance abuse in the past 5 years or other medical illness that might produce neurologic deficit (such as cerebrovascular disease).
5. Use of systemic antibiotics in the previous month.
6. Use of immunomodulators such as interferons.
7. Chronic medication use will be evaluated in a case-by-case basis
8. Patients will be excluded from this protocol if they are judged by the principal investigator as having a significant impairment in their capacity for judgment and reasoning that compromise their ability to make decisions in their best interest.

EXCLUSION CRITERIA FOR RECOVERED, SEROPOSITIVE, OSPA VACCINATED AND HEALTHY VOLUNTEERS CONTROLS:

In addition to the above applicable exclusion criteria (general exclusion criteria and exclusion criteria for PTLDS patients and Lyme arthritis controls), these individuals will be excluded for:

1. Pre-existing or concurrent serious chronic medical or psychiatric illness.

EXCLUSION CRITERIA FOR MULTIPLE SCLEROSIS CONTROLS:

In addition to the above general exclusion criteria, these individuals will be excluded for:

1. Pre-existing or concurrent serious psychiatric or chronic medical illness besides Multiple Sclerosis.
2. Past history of significant head trauma, alcohol or substance abuse in the past 5 years or other medical illness, besides Multiple Sclerosis, that might produce neurologic deficit (such as cerebrovascular disease).
3. Previously received total lymphoid irradiation (TLI) or cladribine.
4. Has used immunoactive medications (excluding beta-interferon) in the three months preceding the study.
5. In the three months prior to the study initiation, was given such investigational treatments as plasmapheresis, hyperbaric oxygen, gangliosides, Copolymer 1, etc.

ELIGIBILITY OF SPECIAL POPULATIONS

Children: Children 13 years and older are eligible to participate in the PTLDS cohort because the condition under study can affect children. This age was selected as appropriate for the children to provide assent to and comply with the study procedures. Children younger than 13 will be excluded from the PTLDS cohort, and no children will be enrolled in the other study cohorts.

Pregnant and lactating women: Pregnant and lactating women are excluded from study participation. An enrolled participant who becomes pregnant during the study will be withdrawn

Adults who lack capacity to consent: Adults who lack decision-making capacity to provide informed consent are excluded at screening, and enrolled adult participants who permanently lose the ability to consent during study participation will be withdrawn

NIH staff members: NIH staff may be enrolled if they meet eligibility criteria. Neither participation nor refusal to participate as a subject in the research will have an effect, either beneficial or adverse, on the participant s employment or position at NIH. Every effort will be made to protect participant information, but such information may be available in medical records and may be available to authorized users outside of the study team in both an identifiable and unidentifiable manner.

Ages: 13 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Primary clinical
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 1996-06-13 (Actual)

PRIMARY OUTCOMES:
Assemble and follow a well-characterized cohort of patients with post-treatment Lyme disease syndrome and relevant controls | duration of the study
  This protocol serves as the basis for multiple parallel lines of investigation in different aspects of Lyme disease and PTLDS. The formation of the cohort and follow up are the main outcomes.

SECONDARY OUTCOMES:
Explore biological markers of B. burgdorferi infection and PTLDS | duration of study
  Explore biological market of B. burgdorferi infection and PTLDS
Development of new tests for Lyme disease and PTLDS | duration of study
  Development of new tests for Lyme disease and PTLDS
Assessment of the immunological response in patients with PTLDS | duration of study
  Assessment of the immunological response in patients with PTLDS
Assessment of clinical course and outcomes of patients with PTLDS | duration of study
  Assessment of clinical course and outcomes of patients with PTLDS

CONTACTS AND LOCATIONS:
Overall Officials: Adriana R Marques, M.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if the research results will reveal a need to disclose IPD, therefore it is undecided if we plan to make IPD available.

REFERENCES:
- [Derived] Marques AR, Yang X, Smith AA, Zhuang X, Turk SP, Williams CD, Law MA, Barbour AG, Pal U. Citrate Anticoagulant Improves the Sensitivity of Borreliella (Borrelia) burgdorferi Plasma Culture. J Clin Microbiol. 2017 Nov;55(11):3297-3299. doi: 10.1128/JCM.01046-17. Epub 2017 Sep 6. No abstract available. PMID 28878005
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_1996-I-0052.html